CLINICAL TRIAL: NCT00001718
Title: Facilitation of Oral Bolus Propulsion Using Electropalatography in Patients With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980135; 98-CC-0135
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-07

CONDITIONS: Deglutition Disorders; Dysphagia
Keywords: Biofeedback; Swallowing; Swallowing Therapy; Tongue/Palate; Ultrasound; Dysphagia
MeSH Terms: conditions — Deglutition Disorders

INTERVENTIONS:
Device: Electropalatography

SUMMARY:
Electropalatography (EPG), a noninvasive device that provides specific visual output on tongue-palate contact, has well-established usefulness as a biofeedback tool in speech therapy. While EPG has also been shown to be capable of revealing the details of linguopalatal interactions during swallowing, its applicability in swallowing therapy has not been evaluated to date. This study will determine if EPG can facilitate bolus propulsion in patients presenting with swallowing problems of the oral phase. Seven patients with oral dysphagia will be selected to serve as subjects based on specific inclusion and exclusion criteria, and each will be custom-fitted with a pseudo-palate. Each patient will undergo four 45-minute sessions of biofeedback training with emphasis on developing systematic front-to-back anchoring of the tongue against the palate during propulsion of liquid and semisolid boluses. Ultrasound imaging will be used to determine swallow durations and identify oral deficits of swallowing before the EPG biofeedback training, and to identify any changes that may result from the training. Quantitative measurements will also be made of the swallow-related EPG contact timing and pattern before and after training and compared for each individual subject as a function of training and bolus volume. Appropriate statistical analyses will be conducted.

DETAILED DESCRIPTION:
Electropalatography (EPG), a noninvasive device that provides specific visual output on tongue-palate contact, has well-established usefulness as a biofeedback tool in speech therapy. While EPG has also been shown to be capable of revealing the details of linguopalatal interactions during swallowing, its applicability in swallowing therapy has not been evaluated to date. This study will determine if EPG can facilitate bolus propulsion in patients presenting with swallowing problems of the oral phase. Ten patients with oral dysphagia will be selected to serve as subjects based on specific inclusion and exclusion criteria, and each will be custom-fitted with a pseudo-palate. Each patient will undergo four 45-minute sessions of biofeedback training with emphasis on developing systematic front-to-back anchoring of the tongue against the palate during propulsion of liquid and semisolid boluses. Ultrasound imaging will be used to determine swallow durations and identify oral deficits of swallowing before the EPG biofeedback training, and to identify any changes that may result from the training. Quantitative measurements will also be made of the swallow-related EPG contact timing and pattern before and after training and compared for each individual subject as a function of training and bolus volume. Appropriate statistical analyses will be conducted.

ELIGIBILITY:
Patients who have undergone comprehensive swallowing evaluations (i.e., ultrasound and/or videofluoroscopic swallow studies, oral sensorimotor examination, and swallowing questionnaire) in the Speech Pathology Section and have been found to have dysphagia with prominent oral signs.

All subjects must be alert and oriented to time and place, able to ingest food by mouth, and have intact or aided hearing and vision.

No patients that exhibit oral apraxia, dementia, aphasia, behavioral problems, and endentousness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 1998-07; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Chi-Fishman G, Stone M. A new application for electropalatography: swallowing. Dysphagia. 1996 Fall;11(4):239-47. doi: 10.1007/BF00265208. PMID 8870350
- [Background] Chi-Fishman G, Stone M, McCall GN. Lingual action in normal sequential swallowing. J Speech Lang Hear Res. 1998 Aug;41(4):771-85. doi: 10.1044/jslhr.4104.771. PMID 9712125
- [Background] Logemann JA, Kahrilas PJ, Hurst P, Davis J, Krugler C. Effects of intraoral prosthetics on swallowing in patients with oral cancer. Dysphagia. 1989;4(2):118-20. doi: 10.1007/BF02407156. PMID 2701094